CLINICAL TRIAL: NCT01040871
Title: A Randomized, Open-Label, Multicenter Phase 2 Study of the Combination of VELCADE, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With Newly Diagnosed Non-Germinal Center B-Cell Subtype of Diffuse Large B-Cell Lymphoma
Brief Title: Study of the Combination of VELCADE, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone in Patients With Newly Diagnosed Non-Germinal Center B-Cell Subtype of Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Collaborators: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 26866138-LYM-2034; NCT01826084 (obsolete NCT alias)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Results first posted 2013-11-27 (Estimated); Last update posted 2014-01-13 (Estimated); Status verified 2013-12

CONDITIONS: Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — Bortezomib; Rituximab; Cyclophosphamide; Doxorubicin; Prednisone; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- VR-CAP (Experimental): VR-CAP arm received rituximab 375 mg/m2 IV on Day 1, cyclophosphamide 750 mg/m2 IV on Day 1, doxorubicin 50 mg/m2 IV on Day 1, VELCADE 1.3 mg/m2 IV on Days 1, 4, 8, and 11, and prednisone 100 mg/m2 orally on Days 1 through 5 of each 21-day (3-week) cycle for up to 6 cycles.
  Interventions: Drug: VELCADE; Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone
- R-CHOP (Active Comparator): R-CHOP received rituximab 375 mg/m2IV on Day 1, cyclophosphamide 750 mg/m2 IV on Day 1, doxorubicin 50 mg/m2 IV on Day 1, vincristine 1.4 mg/m2 (maximum total of 2 mg) IV on Day 1, and prednisone 100 mg/m2 orally on Days 1 through 5 of each 21-day (3-week) cycle for up to 6 cycles.Prednisone
  Interventions: Drug: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Prednisone; Drug: Vincristine

INTERVENTIONS:
Drug: VELCADE — VELCADE intravenous on Days 1, 4, 8, and 11 of a 21 day (3 week) cycle for 6 cycles.
  Arms: VR-CAP
Drug: Rituximab — Rituximab intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles
Drug: Cyclophosphamide — Intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles
Drug: Doxorubicin — Intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles
Drug: Prednisone — Orally on Day 1 to Day 5 of a 21 day (3 week) cycle for 6 cycles
Drug: Vincristine — Intravenous on Day 1 of a 21 day (3 week) cycle for 6 cycles
  Arms: R-CHOP

SUMMARY:
This is a randomized, open-label, active-control, parallel-group, multicenter, multinational Phase 2 Study of the efficacy and safety of VELCADE, Rituximab, Cyclophosphamide, Doxorubicin, and Prednisone (VR-CAP) or Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, and Prednisone (R-CHOP) in Patients With Newly Diagnosed Non-Germinal Center B-Cell (non-GCB) Subtype of Diffuse Large B-Cell Lymphoma (DLBCL)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years or older.
* Newly Diagnosed non-GCB subtype of DLBCL (Stage II, III or IV).
* At least 1 measurable site of disease.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Female subjects must be postmenopausal (for at least 6 months), surgically sterile, abstinent, or, if sexually active, be practicing an effective method of birth control before entry and throughout the study; and have a negative pregnancy test at screening.
* Male subjects must agree to use a double barrier method of birth control

Exclusion Criteria:

* Prior treatment with VELCADE.
* Prior extended radiotherapy or chemotherapy for lymphoma
* More than 150 mg/m2 of prior doxorubicin
* Major surgery within 3 weeks of study.
* Peripheral neuropathy or neuralgia of Grade 2 or worse.
* Active CNS lymphoma
* Diagnosed or treated for a malignancy other than NHL, with some exceptions
* Pregnant or breast feeding
* Active systemic infection
* Documented of suspected human immunodeficiency virus (HIV)/AIDS
* Uncontrolled or severe cardiovascular disease
* Known allergies, hypersensitivity or intolerance to study drugs
* Serious medical condition that could interfere with study
* Concurrent treatment with another investigational agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2010-01; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Millennium Pharmaceuticals, Inc.
Locations (1):
- Universitair Ziekenhuis Gent - UZ GENT, Hematologie, 9K12IE 9de verdiep- polikliniek Hematologie, Ghent, Belgium

REFERENCES:
- [Derived] Offner F, Samoilova O, Osmanov E, Eom HS, Topp MS, Raposo J, Pavlov V, Ricci D, Chaturvedi S, Zhu E, van de Velde H, Enny C, Rizo A, Ferhanoglu B. Frontline rituximab, cyclophosphamide, doxorubicin, and prednisone with bortezomib (VR-CAP) or vincristine (R-CHOP) for non-GCB DLBCL. Blood. 2015 Oct 15;126(16):1893-901. doi: 10.1182/blood-2015-03-632430. Epub 2015 Jul 31. PMID 26232170

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 164 participants were randomized, three participants did not receive study treatment (2 in the VR-CAP and 1 in the R-CHOP arm) for a total of 161 treated.
Period: Overall Study
Arm/Group | VR-CAP | R-CHOP
Started | 84 (Intent to Treat, Randomized) | 80 (Intent to Treat, Randomized)
Completed | 71 | 73
Not Completed | 13 | 7
Not completed — Adverse Event | 6 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Death | 1 | 3
Not completed — Lack of Efficacy | 1 | 1
Not completed — drug supply issue | 1 | 0
Not completed — Randomized and Not Treated | 2 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat, Randomized
Groups:
- VR-CAP: VELCADE, Rituximab, Cyclophosphamide, Doxorubicin and Prednisone
- R-CHOP: Rituximab, Cyclophosphamide, Doxorubicin, Vincristine and Prednisone
- Total: Total of all reporting groups
Arm/Group | VR-CAP | R-CHOP | Total
Number analyzed (Participants) | 84 | 80 | 164
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (15.00) | 57.8 (13.83) | 57.2 (14.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 43 | 33 | 76
  Male | 41 | 47 | 88
Region of Enrollment [Number; unit: participants]
  Russian Federation | 22 | 14 | 36
  Turkey | 4 | 12 | 16
  Korea, Republic of | 6 | 6 | 12
  Malaysia | 5 | 3 | 8
  Canada | 3 | 3 | 6
  India | 2 | 4 | 6
  Brazil | 2 | 3 | 5
  Argentina | 2 | 1 | 3
  Singapore | 2 | 1 | 3
  Mexico | 0 | 1 | 1
  Germany | 13 | 8 | 21
  Portugal | 5 | 7 | 12
  Italy | 2 | 6 | 8
  Czech Republic | 3 | 4 | 7
  Spain | 5 | 2 | 7
  France | 2 | 4 | 6
  Belgium | 4 | 1 | 5
  Ireland | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate
Description: Complete response was evaluated by an Independent Radiology Review Committee using available computed tomography (CT) and positron emission tomography (PET) scans collected at Baseline, end of cycle 3, and end of cycle 6 (or end of treatment) based on the Revised Response Criteria for Malignant Lymphoma.
  1. Complete disappearance of all detectable clinical evidence of disease and disease-related symptoms if present before therapy.
  2. PET scan was negative.
  3. The spleen and/or liver, if enlarged before therapy on the basis of physical examination or CT scan, was not palpable on physical examination and was considered normal size by imaging studies; all splenic and hepatic nodules related to lymphomas disappeared.
  4. If bone marrow was involved before treatment, the infiltrate cleared on repeated bone marrow biopsy.
  5. No new sites of disease were detected.
Time Frame: 6 cycles
Population: All randomized subjects with non-GCB DLBCL who received at least 1 dose of any study drug, had at least 1 measurable lesion at baseline, and had at least 1 post-baseline response assessment
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 76 | 74
percentage of participants | 64.5 [55.4 to 73.5] | 63.5 [54.3 to 72.7]
Statistical Analysis 1: Comparison: VR-CAP vs R-CHOP; Test type: Superiority or Other; p = 0.915, Cochran-Mantel-Haenszel; Stratified by IPI score; Odds Ratio (OR) = 1.038, 95% CI 2-sided [0.529 to 2.037] — Odds ratio: VR-CAP CR rate relative to R-CHOP CR rate

2. Secondary Outcome: Overall Response Rate
Description: Overall response = Complete Response (CR) + Partial Response (PR) Response was evaluated by an Independent Radiology Review Committee using available computed tomography (CT) and positron emission tomography (PET) scans collected at Baseline, end of cycle 3, and end of cycle 6 (or end of treatment) based on the Revised Response Criteria for Malignant Lymphoma.
  Complete Response: see primary endpoint Partial Response: At least a 50% decrease in the sum of the product of the diameters (SPD) of up to 6 of the largest dominant nodes or nodal masses.
Time Frame: 6 cycles
Population: as for outcome 1
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 76 | 74
percentage of participants | 93.4 [88.7 to 98.1] | 98.6 [96.4 to 100.0]

3. Secondary Outcome: Rate of Durable Response
Description: Proportion of subjects who achieved a CR or PR with duration of at least 6 months. Duration of response (CR or PR) was calculated from the date of initial documentation of a response to the date of first documented evidence of disease progression or death due to disease progression. Response was evaluated by an Independent Radiology Review Committee using available computed tomography (CT) and positron emission tomography (PET) scans collected at Baseline, end of cycle 3, end of cycle 6 (or end of treatment) based on the Revised Response Criteria for Malignant Lymphoma.
Time Frame: Median follow up approx. 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 76 | 74
percentage of participants | 53.9 [44.5 to 63.4] | 67.6 [58.6 to 76.5]

4. Secondary Outcome: Rate of Durable Complete Response
Description: Proportion of subjects who achieved a CR with duration of at least 6 months
Time Frame: Median follow up approx 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 76 | 74
percentage of participants | 44.7 [35.3 to 54.1] | 47.3 [37.7 to 56.9]

5. Secondary Outcome: Subsequent Anti-lymphoma Therapy Rate at 1-year
Description: Kaplan-meier estimate of subsequent anti-lymphoma therapy at 1-year. Time to subsequent anti-lymphoma therapy was measured from the date of randomization to the start date of new treatment. Death due to disease progression prior to subsequent therapy was considered as an event. Otherwise, time to next anti-lymphoma treatment was censored at the date of death or the last date known to be alive.
Time Frame: 1 year
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 84 | 80
percentage of participants | 71.1 [57.9 to 80.8] | 80.2 [68.8 to 87.9]

6. Secondary Outcome: Progression-free Survival (PFS)Rate at 1-year
Description: Kaplan-meier estimate of progression-free survival at 1-year. Progression-free survival was defined as the interval between the date of randomization and the date of first documented evidence of disease progression or death.
Time Frame: 1 year
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of partipants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 84 | 80
percentage of partipants | 78.9 [67.2 to 86.8] | 83.9 [72.7 to 90.8]

7. Secondary Outcome: Overall Survival Rate at 1-year
Description: Kaplan-meier estimate of overall survival at 1-year measured from date of randomization.
Time Frame: 1 year
Population: Intent to Treat Population
Measure: Number (95% Confidence Interval); unit: percentage of partipants
Arm/Group | VR-CAP | R-CHOP
Number analyzed (Participants) | 84 | 80
percentage of partipants | 94.1 [84.6 to 97.8] | 84.2 [73.2 to 91.0]

8. Secondary Outcome: Change in Fatigue and Patient Utility Scores
Time Frame: 18-24 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: Number at risk is based on the safety population defined as patients who were randomized and received at least one dose of study drug. A total of 164 participants were randomized and 3 participants did not receive study treatment (2 in the VR-CAP arm, 1 in the R-CHOP arm) for a total of 161 treated (82 in the VR-CAP arm, 79 in the R-CHOP arm).
Arm/Group | VR-CAP | R-CHOP
Serious Adverse Events (participants affected / at risk) | 31/82 | 27/79
Other Adverse Events (participants affected / at risk) | 73/82 | 72/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | VR-CAP (N=82) | R-CHOP (N=79)
Febrile neutropenia (Blood and lymphatic system disorders) | 7 | 7
Neutropenia (Blood and lymphatic system disorders) | 4 | 5
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 4 | 3
Device related infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 1 | 1
Lung infection (Infections and infestations) | 2 | 0
Septic shock (Infections and infestations) | 1 | 1
Abscess neck (Infections and infestations) | 0 | 1
Hepatitis viral (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Oral candidiasis (Infections and infestations) | 1 | 0
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Dyphagia (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pyrexia (General disorders) | 5 | 0
Asthenia (General disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 1 | 0
Malaise (General disorders) | 1 | 0
Performance status decreased (General disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Arrhythmia (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Extrasystoles (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1
Hypertension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 2 | 0
Hyperphosphatasaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
International normalised ratio increased (Investigations) | 0 | 1
Skin discoloration (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | VR-CAP (N=82) | R-CHOP (N=79)
Constipation (Gastrointestinal disorders) | 24 | 25
Dyspepsia (Gastrointestinal disorders) | 11 | 7
Stomatitis (Gastrointestinal disorders) | 9 | 7
Abdominal pain upper (Gastrointestinal disorders) | 9 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 23 | 15
Headache (Nervous system disorders) | 9 | 8
Hypoaesthesia (Nervous system disorders) | 8 | 4
Neuralgia (Nervous system disorders) | 9 | 0
Dysgeusia (Nervous system disorders) | 5 | 1
Fatigue (General disorders) | 21 | 11
Oedema peripheral (General disorders) | 14 | 5
Chills (General disorders) | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 3
Nasopharyngitis (Infections and infestations) | 6 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 4
Pruritis (Skin and subcutaneous tissue disorders) | 6 | 1
Anaemia (Blood and lymphatic system disorders) | 19 | 17
Decreased appetite (Metabolism and nutrition disorders) | 13 | 5
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 4
Insomnia (Psychiatric disorders) | 10 | 6
Hepatic function abnormal (Hepatobiliary disorders) | 8 | 9
Conjunctivitis (Eye disorders) | 5 | 1
Weight decreased (Investigations) | 6 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No